CLINICAL TRIAL: NCT03030508
Title: Discovery and Validate of Multi-genetic Biomarkers for Capecitabine in Chinese Colorectal Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Minhang Central Hospital (Other); Xuzhou Medical University (Other); The 97 Hospital of chinese PLA (Unknown); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wansheng Chen, Professor, Director of Department of Pharmacy, Shanghai Changzheng Hospital
Other Study IDs: WChen
Record Dates: First submitted 2017-01-13; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer; Capecitabine
Keywords: biomarks; colorectal cancer; capecitabine; gene polymorphism
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue,blood,urine and stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group cap: Patients receiving capecitabine chemotherapy after operation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
At present, chemotherapy is widely used in the adjuvant treatment of colorectal cancer patients after surgery. Capecitabine is one of the main chemotherapeutic drugs. But the effect is not good enough, the adverse reaction is serious, and the individual differences were significant. The present study shows that these problems are related to the differences in the exposure of capecitabine and its metabolites in different patients. The genetic biomarkers for capecitabine include DRD, MTHFR and TYMS. Mutations in these genes directly affect the expression of metabolic enzymes involved in capecitabine and control the concentration of capecitabine and its metabolites. However, these markers have been obtained through clinical trials in the United States, and their role in predicting the effectiveness or safety of capecitabine and its metabolites has not been validated in Chinese cancer patients.The study was based on a case study of patients with colorectal cancer in China, and capecitabine as the primary postoperative chemotherapy regimen to verify whether the available biomarkers can be used to predict the effectiveness and safety of capecitabine. To clarify the effect of capecitabine on endogenous metabolites, and to study the mechanism of its effect, so as to discover new biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. more than 18 years old;
2. patients with colon cancer diagnosed by biopsy (regardless of cancer stage);
3. received postoperative containing capecitabine chemotherapy;
4. volunteer to participate in the experiment

Exclusion Criteria:

1. pregnant and lactating women;
2. patients with hypersensitivity to fluorouracil or severe metabolic failure;
3. patients with severe infection;
4. patients with other cancers other than colorectal cancer within the first five years of colorectal cancer surgery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients with colorectal cancer receiving first chemotherapy after surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | during chemotherapy
  Adverse Events That Are Related to Treatment
Disease-free survival | Three year disease-free survival

SECONDARY OUTCOMES:
Three year disease free survival rate | Three year disease free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Wansheng Chen, PhD, Study Chair — Department of medicine of Shanghai Changzheng Hospital
Locations (1):
- Department of medicine of Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Sun B, Lu Z. Evaluation of clinical value of single nucleotide polymorphisms of dihydropyrimidine dehydrogenase gene to predict 5-fluorouracil toxicity in 60 colorectal cancer patients in China. Int J Med Sci. 2013 May 20;10(7):894-902. doi: 10.7150/ijms.5556. Print 2013. PMID 23781135
- [Background] Li F, Qin X, Chen H, Qiu L, Guo Y, Liu H, Chen G, Song G, Wang X, Li F, Guo S, Wang B, Li Z. Lipid profiling for early diagnosis and progression of colorectal cancer using direct-infusion electrospray ionization Fourier transform ion cyclotron resonance mass spectrometry. Rapid Commun Mass Spectrom. 2013 Jan 15;27(1):24-34. doi: 10.1002/rcm.6420. PMID 23239314
- [Background] Ikeda K, Oike Y, Shimizu T, Taguchi R. Global analysis of triacylglycerols including oxidized molecular species by reverse-phase high resolution LC/ESI-QTOF MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Sep 1;877(25):2639-47. doi: 10.1016/j.jchromb.2009.03.047. Epub 2009 Apr 7. PMID 19481987
- [Background] Denkert C, Bucher E, Hilvo M, Salek R, Oresic M, Griffin J, Brockmoller S, Klauschen F, Loibl S, Barupal DK, Budczies J, Iljin K, Nekljudova V, Fiehn O. Metabolomics of human breast cancer: new approaches for tumor typing and biomarker discovery. Genome Med. 2012 Apr 30;4(4):37. doi: 10.1186/gm336. PMID 22546809
- [Background] Wu CW, Ng SS, Dong YJ, Ng SC, Leung WW, Lee CW, Wong YN, Chan FK, Yu J, Sung JJ. Detection of miR-92a and miR-21 in stool samples as potential screening biomarkers for colorectal cancer and polyps. Gut. 2012 May;61(5):739-45. doi: 10.1136/gut.2011.239236. Epub 2011 Sep 19. PMID 21930727
- [Background] Deenen MJ, Meulendijks D, Cats A, Sechterberger MK, Severens JL, Boot H, Smits PH, Rosing H, Mandigers CM, Soesan M, Beijnen JH, Schellens JH. Upfront Genotyping of DPYD*2A to Individualize Fluoropyrimidine Therapy: A Safety and Cost Analysis. J Clin Oncol. 2016 Jan 20;34(3):227-34. doi: 10.1200/JCO.2015.63.1325. Epub 2015 Nov 16. PMID 26573078
- [Background] Huang L, Chen F, Chen Y, Yang X, Xu S, Ge S, Fu S, Chao T, Yu Q, Liao X, Hu G, Zhang P, Yuan X. Thymidine phosphorylase gene variant, platelet counts and survival in gastrointestinal cancer patients treated by fluoropyrimidines. Sci Rep. 2014 Jul 16;4:5697. doi: 10.1038/srep05697. PMID 25027354
- [Derived] Li M, Yan T, Chen J, Wang Z, Gao S, Deng Y, Qiu S, Liu X, Huang L, Hou X, Tao X, Yang M, Chen W. Plasma endogenous metabolome as superior biomarkers for adverse effects compared to drug and its metabolites. Future Oncol. 2026 Jan;22(2):167-180. doi: 10.1080/14796694.2025.2609305. Epub 2025 Dec 30. PMID 41468321
- [Derived] Xu J, Lin Z, Chen J, Zhang J, Li W, Zhang R, Xing J, Ye Z, Liu X, Gao Q, Chen X, Zhai J, Yao H, Li M, Wei H. Milk and Egg Are Risk Factors for Adverse Effects of Capecitabine-Based Chemotherapy in Chinese Colorectal Cancer Patients. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221105485. doi: 10.1177/15347354221105485. PMID 35686441
- [Derived] Li M, Sun X, Yao H, Chen W, Zhang F, Gao S, Zou X, Chen J, Qiu S, Wei H, Hu Z, Chen W. Genomic methylation variations predict the susceptibility of six chemotherapy related adverse effects and cancer development for Chinese colorectal cancer patients. Toxicol Appl Pharmacol. 2021 Sep 15;427:115657. doi: 10.1016/j.taap.2021.115657. Epub 2021 Jul 29. PMID 34332992
- [Derived] Li M, Chen J, Deng Y, Yan T, Gu H, Zhou Y, Yao H, Wei H, Chen W. Risk prediction models based on hematological/body parameters for chemotherapy-induced adverse effects in Chinese colorectal cancer patients. Support Care Cancer. 2021 Dec;29(12):7931-7947. doi: 10.1007/s00520-021-06337-z. Epub 2021 Jul 2. PMID 34213641